CLINICAL TRIAL: NCT00680004
Title: The Value of Dynamic CTA During the Follow-up of EndoVascular Aortic Replacement (EVAR): a Pilot Study
Brief Title: Dynamic Computed Tomography Angiography (CTA) Follow-up for EndoVascular Aortic Replacement (EVAR)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Professor Leo Schultze Kool, UMC St Radboud Nijmegen
Other Study IDs: dCTA-2006-YH
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2008-05

CONDITIONS: Aortic Aneurysm
Keywords: Dynamic CTA; follow-up; EVAR
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Preoperative patients planned for a CT prior to an endograft implantation procedure
- 2: Patients who underwent a complicated endograft implant and/or with increased risk of complications

SUMMARY:
This pilot study aims to quantitatively characterize the stresses and forces on an implanted endograft during the cardiac cycle in patients scheduled for standard endograft follow-up. The developed techniques will be applied in future studies for characterizing and comparing the currently commercially available endografts so as to gain insight into the mechanisms underlying potential endograft failure. In addition, to assist in developing endografts with long-term durability and functioning characteristics for the benefit of the patient

DETAILED DESCRIPTION:
Endovascular Aortic replacement (EVAR) for the treatment of aortic aneurysms in patients at risk of aneurysm rupture is an established endovascular technique (ref: Blankensteijn, NEJM, 2005). However, the development of the endograft design is ongoing in order to prevent late endograft failure (e.g. graft breakage, graft displacement). The stresses and forces applied to the endograft by the high physiological forces and stresses in the aorta have an effect on the durability and functioning of the endograft. The stresses and forces that occur during movement may be reflected by movement of the endograft itself during the cardiac cycle. Standard patient follow-up involves transverse CT imaging to detect endograft leakage. However, transverse imaging does not provide information on endograft displacement but does provide information on shrinkage of the aneurysm after endograft placement. Therefore, additional information on the longitudinal displacement of the endograft during the cardiac cycle may assist in determining the optimal characteristics of a durable endograft and therefore benefit the patient in the long-term. Evaluation of the stresses and forces by calculating longitudinal displacement of the endograft appears possible by applying a cardiac CT technique, namely, dynamic CTA (computed tomography angiography), on an endovascular device. To our knowledge, this new approach will yield new in vivo data on endograft behavior.

This pilot study aims to quantitatively characterize the stresses and forces on an implanted endograft during the cardiac cycle in patients scheduled for standard endograft follow-up. In addition, in order to have the possibility to compare the movement of the aorta pre- and post-endograft placement, the aorta of patients planned for an endograft implantation procedure and who are thus already planned to undergo a clinical CT will also instead be scanned using ECG gated dynamic CTprotocol.

The developed techniques will be applied in future studies for characterizing and comparing the currently commercially available endografts so as to gain insight into the mechanisms underlying potential endograft failure, and in addition, to assist in developing endografts with long-term durability and functioning characteristics for the benefit of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative patients planned for a CT prior to an endograft implantation procedure
* Patients who underwent a complicated endograft implant and/or with increased risk of complications
* 18 years of age or older
* Patients who have given their informed consent

Exclusion Criteria:

* Known allergy for contrast medium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing either a preoperative CT procedure or with an implanted aortic endoprothesis (-graft) presenting to the department of radiology for a scheduled follow-up CTA procedure.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-09 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
to quantitatively characterize the stresses and forces on an implanted endograft during the cardiac cycle in terms of longitudinal movement

SECONDARY OUTCOMES:
evaluate the integrity of the endograft by visualization using CT in the longitudinal and transversal plane at several moments during the cardiac cycle versus the standard transverse plane method

CONTACTS AND LOCATIONS:
Overall Officials: Leo Schultze Kool, MD, Principal Investigator — UMC St Radboud Nijmegen
Locations (1):
- UMC St Radboud, Nijmegen, Netherlands